CLINICAL TRIAL: NCT03214445
Title: Reparación y Sellado de Restauraciones de Amalgama y Resinas Compuestas Para el Incremento de Su Longevidad Repair and Sealing of Amalgam and Composite Resins to Increase of Longevity
Brief Title: Sealing Defective Margins of Composite Restorations With Fluid Composite Resin Nanofiller Reinforced
Acronym: SEAL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Profesor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012/10
Record Dates: First submitted 2017-05-18; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Dental Caries; Minimally Invasive; Repair
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: prospective, double blind randomized clinical trial under the recommendations of CONSORT. The statistical unit was considered the patient (n=60), with at least 3 composite resins with marginal defects , randomized into 3 groups A=Sealed with flow composite reinforced with nanofiller , B= Sealed with resin sealant , and C=Control, without intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The evaluated restorations will be coded, and the data will be delivered in sealed envelopes without any identification of the patient, the data will be processed without identification of the groups. The sealant and the resin will be the same color so the evaluator will not be able to differentiate the treatments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- resin composite with nanofiller. (Experimental): 30 restorations of resin composite occlusal, molars or premolars, with values of 3 or 4 for the parameter marginal adaptation according to the FDI criteria randomized assigned in this group
  Interventions: Procedure: Sealing margins with flow composite
- sealant based on resin (Active Comparator): 30 restorations of resin composite occlusal, molars or premolars, with values of 3 or 4 for the parameter marginal adaptation according to the FDI criteria randomized assigned in this group
  Interventions: Procedure: Sealing margins with seal
- Control (No Intervention): The restorations were evaluated without treatment about defective restoration that was considered clinically acceptable.

INTERVENTIONS:
Procedure: Sealing margins with flow composite — Seal the margin of restoration with Composite flow with nanofiller
  Arms: resin composite with nanofiller.
Procedure: Sealing margins with seal — Seal the margin of restoration with sealant without filler
  Arms: sealant based on resin

SUMMARY:
the patient (n=60), with at least 3 composite resins with marginal defects , randomized into 3 groups A=Sealed with flow composite reinforced with nanofiller , B= Sealed with resin sealant , and C=Control, without intervention , and then assessed by the FDI criteria for clinical performance and longevity of restorations

DETAILED DESCRIPTION:
This is a prospective, double-blind randomized clinical trial under the recommendations of CONSORT. The statistical unit was considered the patient (n=60), with at least 3 composite resins with marginal defects , randomized into 3 groups A=Sealed with flow composite reinforced with nanofiller , B= Sealed with resin sealant , and C=Control, without intervention.

Inclusion criteria:

* Age 18 or older
* High risk of caries.
* With restorations of resin composite occlusal, molars or premolars, with values of 3 or 4 for the parameter marginal adaptation according to the FDI criteria.

Exclusion criteria:

* Patients with the impossibility of mouth opening or dental treatments.
* Patients with allergies to any of the materials used.
* The presence of adjacent to the restoration or secondary caries.
* Patients with prior sealed of their restorations.

The volunteers were informed of the objectives and risks of treatment, as well as the freedom to leave the study. It explained in detail the clinical procedure which was submitted and proceeded to sign the informed consent according to the rules of the Ethics Committee of the Faculty of Dentistry of the University of Chile.

Then were assigned the sample within 3 groups of randomly with software Eclipse SDK 4.2.1: (1) sealing with fluid composite resin restorations with nano filled and universal adhesive, (2) sealant adhesive based on resin composite resin with universal adhesive and (3) group control or untreated.

Initial examination Examination of patients was performed independently by two calibrated evaluators, in case of disagreement operators were consulted with a third operator, this in a clinical field well lit, with the tooth surface clean with brush of prophylaxis and water, for the clinical examination was used to mirror No 5 (Hu-Friedy Mfg. Co. Inc., Chicago, IL, USA), probe of caries straight with active diameter of 150 μm portion (Deppeler, Swiss Dental) and caries probe straight with active portion of diameter 250 μm (Deppeler, Swiss Dental), both indicated by the FDI. For an optimal value in the parameter of marginal adaptation, the gap should be a size less than or equal to the diameter of the active portion of the probes.

Procedure

Once selected patients and their restorations, were polished using aluminum oxide disks with complete series (Sof-Lex. 3M ESPE) and polished tips (Diacomp, Brasseler).

Each restoration to seal received an identification code, which was awarded randomly belong to an experimental group, as described previously. The tabulation and data of each treatment were conducted in the program Microsoft Excel 2011.

Software Cariogram was used to assess the parameters for the analysis of risk cariogenic: the experience of caries, diseases related, content diet, the frequency of diet, the quantity of plaque, fluor exposition , salivary secretion, capacity buffer and clinical judgment.

Treatment and clinical intervention groups

Group 1::Sealed with fluid resin composite with nanofiller.

Once cleaned the restoration with prophylaxis hard brush and water, at low speed. The procedure was performed under absolute isolation with a rubber dam and using ejector to remove saliva and excess water. Following the protocol of conditionate surface with orthophosphoric acid 35%, for 15 seconds, washed ( abundant water by 30 s) and dried with compressed air from the syringe for 15 s. Then proceeded with the application of adhesive (Single Bond Universal, 3M ESPE) with brush (Microbrush International, Grafton, USA) and friction against the surface for 20 seconds, dried for 5 seconds for evaporation of the solvent remaining and photopolymerized for 10 seconds, using light curing (2500 Curing light, 3M ESPE).

Applied in marginal defects of nanoparticle flowable composite resin (Filtek Flow Z350XT, 3M ESPE) with instrument for cement application of calcium hydroxide (PICH, Hu Friedy Mfg. Co Inc., Chicago, IL, USA), it is polymerized for 20 seconds (2500 Curing light, 3 M ESPE).

The occlusal checked was controlled with paper articulate with 200 microns of width (Bausch Articulating Papers, Inc., USA), occlusal adjustments and wear were carried out with a stone No. 3 high speed (SSWhite, USA).

Group 2: Sealed with sealant based on resin. Once cleaned the restoration with prophylaxis hard brush and water, at low speed. The procedure was performed under absolute isolation with a rubber dam and using ejector to remove saliva and excess water. Following the same Protocol of conditioning, this was done with orthophosphoric acid 35%, for 15 seconds, wash by 30 seconds and dried with compressed air from the syringe for 15 seconds. Then proceeded with the application of adhesive (Single Bond Universal, 3M ESPE) with brush (Microbrush International, Grafton, USA) and friction against the surface for 20 seconds, flow of air for 5 seconds for evaporation of the solvent remaining and polymerizing for 10 seconds, using light curing (2500 Curing light, 3M ESPE).

Applied in marginal defects sealant of pits and fissures based on composite resin (Clinpro Sealant, 3 M ESPE) instrument of cement application of calcium hydroxide (PICH, Hu Friedy Mfg. Co Inc., Chicago, IL, USA), polymerized for 20 seconds (2500 Curing light, 3 M ESPE).

The occlusal checked was controlled with paper articulate 200 microns width (Bausch Articulating Papers, Inc., USA), occlusal adjustments and wear were carried out with stone No. 3 high speed (SSWhite, USA).

Group 3: control. The restorations were evaluated without treatment about defective restoration that was considered clinically acceptable.

Evaluation of treatments

Clinical assessments were made at 6 and 12 months in the parameters marginal adaptation, marginal staining and secondary caries and sealant retention.

Examination was performed independently by two calibrated operators, in case of disagreement were consulted with a third operator, this in a clinical field well lit, with the clean tooth surface with brush of prophylaxis and water, for the clinical examination was used the same methodology and instrumentation that examination.

Analysis of the clinical performance of the treatment groups

To evaluate the behavior of these treatments, after 6 and 12 months, was made the comparison versus baseline, whose valuation assigned to the subsequent application of seal evaluation was 1 (FDI), with the current state of the restoration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* High risk of caries.
* With restorations of resin composite occlusal, molars or premolars, with values of 3 or 4 for the parameter marginal adaptation according to the FDI criteria.

Exclusion Criteria:

* Patients with impossibility of mouth opening or dental treatments.
* Patients with allergies to any of the materials used.
* Presence of adjacent to the restoration or secondary caries.
* Patients with prior sealed of their restorations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Marginal adaptation | 6 month
  ( mm of bridge between tooth and restorations )
Marginal staining, | 4 years
  ( + >50% diameter / - <50% diameter)
Retention of seal ( is present + / was loose -) | 4 years
  Loss of restoration

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martin, Study Director — U de Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez E, Martin J, Vildosola P, Estay J, de Oliveira Junior OB, Gordan V, Mjor I, Gonzalez J, Loguercio AD, Moncada G. Sealing composite with defective margins, good care or over treatment? Results of a 10-year clinical trial. Oper Dent. 2015 Mar-Apr;40(2):144-52. doi: 10.2341/14-143-C. Epub 2014 Dec 23. PMID 25535778